CLINICAL TRIAL: NCT02078596
Title: Double Blind Placebo Controlled Study of Depakote (Divalproex Sodium) in Children With Temper Outbursts and Severe Mood Swings
Brief Title: Depakote (Divalproex Sodium) for Children With Temper Dysregulation and Severe Mood Swings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4592R
Record Dates: First submitted 2014-03-02; First posted 2014-03-05 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Irritable Aggression
Keywords: temper outbursts; pediatric aggression; irritability
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Divalproex (Experimental): Divalproex at 10 mgs/lb
  Interventions: Drug: Divalproex
- Sugar Pill (Placebo Comparator): Equivalent 250 mg pills titrated to 10 mgs / lb over six weeks
  Interventions: Drug: Divalproex

INTERVENTIONS:
Drug: Divalproex — Patients were randomly assigned to receive divalproex or placebo first, follow by the converse treatment, for six weeks each
  Other Names: Divalproex (Depakote)

SUMMARY:
Though the Disruptive Disorders of Childhood and Adolescence are a major source of morbidity and fill a large proportion of special education slots, specific pharmacologic treatment is available only for those children with Attention Deficit/Hyperactivity Disorder. Other disruptive children are usually said to "have" Oppositional Defiant or Conduct Disorder. These diagnoses are useful descriptively but they do not have specific treatment implications In the course of treating adolescents with explosive tempers and severe mood swings with Depakote (divalproex sodium), the investigators learned that younger children manifest symptoms that seemed identical to those constituting the adolescent disorder. They were in special education programs and not responding to psychostimulants.

The investigators systematically collected data on these children using the same screening criteria as in our studies of adolescents. Since Depakote has been used to treat seizures in children for more than twenty years, a great deal was known about its safety profile in the pediatric population. The investigators treated 7 children, age 7-12, whose recurrent temper outbursts and chronic mood lability did not respond to individual/family therapy. After parents signed informed consent and children gave assent, these subjects would receive open label Depakote in doses sufficient to reach a blood level between 50-100 micrograms/ml for six weeks. The family received supportive therapy.

DETAILED DESCRIPTION:
The hypothesis to be tested is whether children below age thirteen with the same symptom cluster targeted in that protocol (explosive temper outbursts and severe mood swings, Explosive Mood Disorder) will show the same response to open label Depakote that the adolescents showed. An addition in this protocol is to see if this hypothesis holds under double blind placebo controlled conditions.

The investigators have now completed open treatment with six children and have found that the same criteria that selected a treatment responsive group of adolescents and adults also worked for five of these six children. The investigators now propose to test these findings under double blind conditions. There is no change in the overall safety profile of the treatment. The only change is the addition of a placebo phase. All children will receive active treatment at some point.

In addition, the investigators hypothesize that the clinical syndrome of temper and irritability will tend to resolve with development and that families will not exhibit bipolarity in first degree relatives but will exhibit temper outbursts. This hypothesis will be studied in a follow-up study.

Data Summary

OPEN TRIAL

Patient Age Dose Acute Outcome Long Term Outcome

1. age 10 1000mgs Good Excellent
2. 12 1000mgs Fair-good Poor (non-compliant
3. 10 1000mgs Excellent Good
4. 9 1000mgs Excellent Very good
5. 12 1000mgs Poor Poor
6. 7 500mgs Excellent Good-excellent 7 11 500 mgs Dropped out after 3 weeks; never took meds Poor

BACKGROUND The disruptive disorders of childhood and adolescence are conduct, oppositional-defiant, and attention deficit hyperactivity disorders. Of these, only the latter has a specific pharmacologic treatment. The other two reliably describe problem behaviors of special education classes, chemical dependency units and family courts but have few treatment implications. In a previous communications, the investigators described adolescent subjects with temper outburst and severe mood swings. The investigators labeled the syndrome Explosive Mood Disorder (EMD) and drafted tentative criteria for temper outburst and irritable mood swings (see Inclusion Criteria for EMD). The goal of this study is to demonstrate that Depakote can help a certain type of problem child, one whose disruptiveness is associated with mood dysregulation.

The investigators hypothesized the subjects' mood dysregulation and aggressive disinhibition to be "limbic" pathology. The limbic system is heavily implicated in behavior and emotion, and work by previous investigators suggested episodic dyscontrol can result from limbic irritability. Since carbamazapine and valproic acid are used in limbic seizures and bipolar spectrum disorders, the investigators predicted subjects would improve on divalproex sodium (Depakote), the enteric coated form of valproic acid. The investigators treated thirteen patients meeting the above criteria criteria with open label divalproex sodium. In all cases, there were strikingly beneficial results, including a sharp decline in the frequency and severity of temper outbursts and the severity of mood swings.

The typical patient would progress from irritation to screaming, door-slamming, property destruction or fighting explosively, i.e., without intermediate steps. When not exploding, the patient's affect and frustration tolerance would fluctuate throughout the day. The mood could be irritable, normal or silly but always unpredictable. The patients had chronic interpersonal difficulties, especially with authority figures, thus serious problems with family, school and work were common. They tended to end up with deviant peers, since others could not tolerate the unpredictable interactions. Though some of patients met criteria for Conduct or Oppositional Defiant Disorder, these diagnoses were too heterogeneous to describe the Depakote responders. Cyclothymia and Bipolar II Disorder did not capture the chronic, maladaptive interactions with peers and authority figures. Intermittent Explosive Disorder missed the above plus the connection to mood dysregulation. Borderline Personality implied a specific type of interpersonal pathology (idealization, devaluation, manipulation) that was not necessarily present.

The closest match the investigators found in the literature to our patients was "Emotionally Unstable Character Disorder" (EUCD). This diagnosis described young adults with extreme irritability, mood swings, chronic maladaptive behaviors, and a clear response to a mood stabilizing agent (lithium carbonate). However, even this diagnosis does not capture the explosiveness which is prominent in the sample of Depakote responders. The investigators therefore decided to use the term Explosive Mood Disorder (EMD) to capture the temper outbursts and the mood lability.

Campbell reported hospitalized conduct disordered children with affective (as opposed to predatory) aggression improvement on lithium and Findling reported similar findings in similar outpatients treated with risperidone. The key feature of irritable mood swings is not directly addressed in these studies. In addition, other studies of childhood aggression in Autism, Tourette Syndrome, Bipolar Disorder and mental deficiency suggest a role for risperidone. Nonetheless, it is still not clear what alternative pharmacological treatments for temper driven by irritable mood swings are available.

The investigators treated ten subjects who met screening criteria for EMD with open label Depakote 1000mgs. Baseline evaluation included a full medical and psychiatric interview, the Structured Clinical Interview for Diagnostic and Statistical Manual of Psychiatry-III-R and a record of the total number of explosions during the previous week and thirty days. The latter estimate was obtained from as many sources as possible. At minimum, the patient and one parent had to each give an estimate. As many other sources as possible were also asked to estimate the lability of the patient's mood during the previous week and thirty days. Each week the same information would be obtained about the previous week and a global assessment made as to whether the patient was unimproved, minimally improved, much improved or very much improved.

Twelve adolescents agreed to participate, and two dropped out before receiving an adequate trial. The other ten adolescents showed clear improvement in mood and number of explosions, with the latter typically declining by 90-100%. All ten adolescent patients were judged at least much improved by the psychiatrist, parents and patient. These results were later replicated under double-blind, placebo controlled conditions.

Teachers and parents approached the investigators with children under the age of 13 and asked us to treat them. The investigators obtained permission to collect open label data on those youngsters. The completion of open-label data has led to the current study.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-11
* Meets Screening Criteria (i.e. "Explosive Mood Disorder") A) An explosive temper as evidenced by four or more outbursts of rage, property destruction or fighting per month on minimal provocation B) Mood lability as evidenced by multiple, daily,distinct, shifts from normal to irritable mood with withdrawn or boisterous behavior, occurring without a clear precipitant C) Duration of at least one year when not treated D)Symptoms result in impairment in two or more areas including: school, the law, family, substance use, peers, work E)Symptoms do not occur only during substance toxicity or withdrawal. F)Symptoms not confined to a single setting or context
* Parent and child willing to consent to study
* Inadequate response to an Adequate trial (8 weeks) of Psychotherapy and/or family therapy

Exclusion Criteria:

* Meets criteria for Pervasive Developmental Disorder or Childhood Schizophrenia
* Seizure or other neurological disturbance
* Pregnancy
* Moderate to severe mental deficiency
* Physical exam or laboratory results with significant abnormalities
* Active suicidal or homicidal ideation or history of suicide attempts
* Use of Barbiturates
* Unequivocal manic or hypomanic episode
* Meets criteria for Attention Deficit Hyperactivity Disorder and has not failed a trial of psychostimulants
* Meets criteria for Major Depression in prepuberty
* Sexually active females who are unwilling to use effective methods of contraception.
* Mitochondrial disease or family history of mitochondrial disease

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 1997-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Response | 6 weeks
  70% reduction in overt aggression (as measured by the Modified Overt Aggression Scale) and in irritability (as measured by the six hostility items of the Hopkins Symptoms Checklist)

SECONDARY OUTCOMES:
Modified Overt Aggression Scale | Baseline and at end of 6 weeks and end of 12 weeks
  Measures the severity and frequency of aggressive outbursts producing a single score theat comes the frequency and severity
Six Hostility Items of the Hopkins Symptom Checklist | Baseline, Week 1 and weekly thereafter for up to 12 weeks
  This is a scale that measures irritability items on a 1-5 scale, yielding a total score of up to 30 for the six items

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States